CLINICAL TRIAL: NCT06248125
Title: Effects of Enriched Parent-Infant Interaction on Health in Early Life
Acronym: BIGMIPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2000035858; 1R21HD113998-01 (NIH)
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Parenting Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Singing intervention (music with enrichment) (Experimental): The goal of this intervention is to improve the frequency and quality of active parent-infant interaction via infant-directed singing. Throughout the 20-week intervention period, parents will be offered a weekly, smartphone- based, music intervention program featuring video-recorded music classes specifically designed for parents with infants. The video classes, which are part of Music Together Wiggle & Sing curriculum, introduce new songs and demonstrate hands-on activities with the songs that parents can easily incorporate into their daily routines. The activities are highly interactive, emphasizing physical contact, gross-motor play, eye contact, cuddling, and rocking. Recordings of these songs will be also provided to supplement parents' learning in the instructional videos with audio-only content (e.g., for parents to use when viewing a video is not convenient). Parents will use the Music Together app and receive a weekly access code for a fresh set of intervention resources.
  Interventions: Behavioral: Singing intervention
- Music listening intervention (music with limited enrichment) (Active Comparator): This intervention follows the same structure as the singing intervention but focuses on the use of passive music listening rather than live singing. On a weekly basis, parents will be provided with a carefully curated music playlist, along with tips on how to effectively incorporate recorded music into their daily lives. These weekly playlists will feature 10 music recordings suitable for everyday scenarios commonly experienced together by parents and infants (e.g., calming lullabies for naptime, exciting play songs for free play). The playlists are intended to serve as background music, thus creating a very different musical experience compared to that of the singing intervention. Each week, parents will receive a link to access a new playlist, along with an information sheet about the music and tips on how to use them. Parents will use Spotify to access the playlists on their smartphones and computers.
  Interventions: Behavioral: Music listening intervention
- Book reading intervention (enrichment with limited music) (Active Comparator): This intervention follows the same structure as the singing intervention, but without the musical elements, while emphasizing enriched parent-infant interaction in non-musical (or less-musical) contexts. Throughout the intervention period, parents will be provided with developmentally appropriate books, carefully selected to encourage increased parent interaction. Along with each book, a demonstration video analogous to the Wiggle and Sing videos used in the singing intervention will be offered. These videos demonstrate techniques to create a rich listening experience for young infants, such as using infant-directed speech and highlighting aspects of illustrations to engage the infant. In line with the singing intervention, the activities will be highly interactive, emphasizing the use of infant-directed speech and physical interactions with their infants.
  Interventions: Behavioral: Book reading intervention
- No intervention (No Intervention): No intervention will be provided.

INTERVENTIONS:
Behavioral: Singing intervention — The goal of this intervention is to improve the frequency and quality of active parent-infant interaction via infant-directed singing.
  Arms: Singing intervention (music with enrichment)
Behavioral: Music listening intervention — This intervention follows the same structure as the singing intervention but focuses on the use of passive music listening rather than live singing.
  Arms: Music listening intervention (music with limited enrichment)
Behavioral: Book reading intervention — This intervention follows the same structure as the singing intervention, but without the musical elements, while emphasizing enriched parent- infant interaction in non-musical (or less-musical) contexts.
  Arms: Book reading intervention (enrichment with limited music)

SUMMARY:
Early life experiences, such as those associated with stable attachment, supportive relationships, and nurturing environments, have profound effects on lifelong physical and mental health. However, children have very different levels of access to such experiences, depending on their family characteristics and associated risk and resilience factors. Low-cost interventions aimed at improving infant environments offer a promising avenue for reducing inequality in early experiences because they require minimal effort to implement. Previous work from the Music lab showed the promise of infant-directed vocalizations, especially music, for enriching parent-infant interaction. Such behaviors are cross-culturally universal, appear regularly in the context of infant care, and have robust effects on infant psychophysiology. In recently completed pilot work, it was found that a brief smartphone-based music intervention achieved high adherence and low attrition; led parents to increase their use of music in soothing their fussy infants; and improved infant mood, as reported via ecological momentary assessment (EMA). Together, these findings show the potential for enriched parent-infant interaction, particularly via infant-directed singing, to improve infant and parent health. Here, a Phase II randomized trial is proposed to explore such effects. Parent/infant dyads (N = 192, infant starting ages 0 to 4 months) will be randomly assigned to one of four conditions: (1) music with enrichment, where parents receive a smartphone-based intervention to learn to sing interactively with their infants, via the early childhood music program Music Together; (2) music with limited enrichment, where parents receive music recordings to listen to with their infants, but are not provided with enrichment activities; (3) enrichment with limited music, where parents receive books to read interactively with their infants, but are not provided with music activities; or (4) a no-treatment control. Throughout the 8-month study, a text-message-based EMA and a survey battery will be used to measure key health outcomes for both infants (distress and recovery, sleep quality, and mood) and parents (mood, mental health status, and parenting efficacy); potential moderators of such effects (demographics, family contextual factors, parent/infant attachment, and infant temperament); as well as parents' degree of engagement in the interventions. Effects will be analyzed both across the intervention groups and relative to the no-treatment control to determine the relative effects of each intervention. The results of this work will determine the effects of low-cost, low-effort early enrichment interventions on basic, everyday health outcomes for infants and parents, test the feasibility of app-based interventions and data collection tools (including in socio-economically disadvantaged families), and provide rich data on the daily lives (including mood, temperament, and sleep variables) of families with young infants. The findings will have particular relevance for underprivileged families and first-time parents, and will set the stage for larger-scale studies of early parent-infant enrichment.

ELIGIBILITY:
Inclusion Criteria:

Investigators will recruit parents or primary caregivers:

* who are the infant's primary caregiver at least 50% of the time during a typical week
* who can communicate and complete surveys in English
* who have a smartphone
* whose infants are healthy.

Exclusion Criteria:

* Investigators will not restrict recruitment of caregivers by age, sex, or any other demographic characteristic.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Infant Mood | post intervention (week 25-26)
  Infant mood measured by a pictorial scale from used in pilot work, measured via Ecological Momentary Assessment (EMA) self-report
Infant Mood | week 31-32
  Infant mood measured by a pictorial scale from used in pilot work, measured via Ecological Momentary Assessment (EMA) self-report
Parent Mood | post intervention (week 25-26)
  Parent mood measured by self-assessed valence, impact, and rationality; from the 3d Mind Model approach to mental state assessment via Ecological Momentary Assessment (EMA) self-report
Parent Mood | week 31-32
  Parent mood measured by self-assessed valence, impact, and rationality; from the 3d Mind Model approach to mental state assessment via Ecological Momentary Assessment (EMA) self-report
Sleep quality | post intervention (week 25-26)
  Measured by the number of night waking episodes that occurred the previous night, and the estimated duration of each episode assessed using the EMA self-report
Sleep quality | week 31-32
  Measured by the number of night waking episodes that occurred the previous night, and the estimated duration of each episode assessed using the EMA self-report
Infant recovery from distress | post intervention (week 25-26)
  Measured by the number of crying episodes that occurred within 3 hours of an ecological momentary assessment ping, and if so, the estimated duration of each episode, and the estimated time to recover from each episode via EMA self-report
Infant recovery from distress | week 31-32
  Measured by the number of crying episodes that occurred within 3 hours of an ecological momentary assessment ping, and if so, the estimated duration of each episode, and the estimated time to recover from each episode via EMA self-report
Parenting efficacy | post intervention (week 25-26)
  Measured by the Karitane Parenting Confidence Scale. It contains 15 items with a possible range of scores of 0-45. Higher scores indicate the parent is feeling more confident.
Parenting efficacy | week 31-32
  Measured by the Karitane Parenting Confidence Scale. It contains 15 items with a possible range of scores of 0-45. Higher scores indicate the parent is feeling more confident.

SECONDARY OUTCOMES:
Parent well-being- Edinburgh Postnatal Depression Scale | post intervention (week 25-26)
  Measured using the Edinburgh Postnatal Depression Scale. It contains 10 items with total score range of 0-30 with scores 13 and above indicating depressive illness.
Parent well-being- Edinburgh Postnatal Depression Scale | week 31-32
  Measured using the Edinburgh Postnatal Depression Scale. It contains 10 items with total score range of 0-30 with scores 13 and above indicating depressive illness.
Parent well-being- Patient Health Questionnaire (PHQ-9) | post intervention (week 25-26)
  Measured using the Patient Health Questionnaire. Total score range 0-27. Higher scores indicate lower physical and mental wellbeing.
Parent well-being- Patient Health Questionnaire (PHQ-9) | week 31-32
  Measured using the Patient Health Questionnaire. Total score range 0-27. Higher scores indicate lower physical and mental wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Mehr, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be shared upon preprinting and/or publication of the results at the Open Science Framework, Zenodo, and other standard scientific data repositories.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Available indefinitely from the time of publication and/or the posting of a preprint.
Access Criteria: All resources will be open-access.
URL: https://zenodo.org/communities/themusiclab